CLINICAL TRIAL: NCT02433990
Title: Risk Factors for Acquired Cardiovascular Disease in Adults With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Susan Fernandes, Principal Investigator, Stanford University
Other Study IDs: IRB-28847
Record Dates: First submitted 2014-05-13; First posted 2015-05-05 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; Acquired Cardiovascular Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult Congenital Heart Disease: 18 years and older with congenital heart disease

SUMMARY:
This research study is to determine the risk factors for acquired heart disease, in adults with congenital heart disease. This knowledge is important to develop and target ways to prevent or delay the onset of acquired heart disease in adults with congenital heart disease.

DETAILED DESCRIPTION:
Advances in surgical and clinical management of patients with congenital heart disease has made survival to adulthood an expectation. Today there are more than 1 million adult survivors of congenital heart disease, but increasing age brings additional concerns for this patient population. Although the literature remains scarce, existing evidence suggests that inactivity, obesity, diabetes, cancer, and acquired cardiovascular disease may be at least as prevalent in patients with congenital heart disease, if not more so, than in an age-matched general population. Acquired cardiovascular disease is likely to impact substantially on long-term survival and quality of life in these patients with palliated and already fragile hearts. This research study is to determine the risk factors for acquired heart disease, in adults with congenital heart disease. This knowledge is important to develop and target ways to prevent or delay the onset of acquired heart disease in adults with congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female over 18 years of age
* Moderate or Complex Congenital Heart Disease
* Willingness to Consent

Exclusion Criteria:

* Pregnancy
* Surgery within 6 months
* Unrepaired cyanotic heart disease
* Patients with Eisenmenger Syndrome physiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Moderate or Complex Congenital Heart Disease
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2019-08-24 (Actual)

PRIMARY OUTCOMES:
Risk factors for acquired cardiovascular disease in adults with congenital heart disease | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Fernandes, PA-C, LP.D., Principal Investigator — Stanford Hospital
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States